CLINICAL TRIAL: NCT06607003
Title: Phase 1 Study of Induced Blood-Stage Malaria in Healthy Malaria-Naive Adults to Assess the Safety and Infectivity of Plasmodium Vivax Challenge Agent and Evaluate Transmission in Mosquito Feeding Assays
Brief Title: Induced Blood-Stage Malaria in Healthy Malaria-Naive Adults to Assess the Safety and Infectivity of Plasmodium Vivax Challenge Agent and Evaluate Transmission in Mosquito Feeding Assays
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10001970; 001970-I
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01-27

CONDITIONS: Malaria
Keywords: IBSM; Challenge; inoculation; Parasitemia; Mosquito Feeding Assay; Malaria Transmission
MeSH Terms: conditions — Malaria; Parasitemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- P. vivax challenge agent derived from PvHMB-CCE001 Main Arm (Experimental): Up to 50 participants will undergo IBSM to further establish safety of the P. vivax challenge agent derived from PvHMB-CCE001 and evaluate transmission to mosquitoes using feeding assays and assess the host response to P. vivax infection.
  Interventions: Biological: P. vivax challenge agent derived from PvHMB-CCE001
- P. vivax challenge agent derived from PvHMB-CCE001 Pilot Arm (Experimental): 2 participants will undergo IBSM to establish the safety and infectivity of the P. vivax challenge agent derived from PvHMB-CCE001.
  Interventions: Biological: P. vivax challenge agent derived from PvHMB-CCE001

INTERVENTIONS:
Biological: P. vivax challenge agent derived from PvHMB-CCE001 — P. vivax challenge agent derived from PvHMB-CCE001 consists of infected and uninfected erythrocytes stabilized in glycerolyte. Challenge agent derived from this bank consists of thawed, washed, infected and uninfected erythrocytes suspended in injectable-grade normal saline.

SUMMARY:
Background:

Malaria is a disease caused by parasites transmitted to people by mosquitoes. Around the world, there were 241 million cases and 627,000 deaths from malaria in 2020. Researchers are working to develop vaccines and treatments for this disease.

Objective:

To learn how malaria develops in people; how the body's immune system reacts to malaria; and how malaria spreads from people to mosquitoes.

Eligibility:

Healthy people in the Washington DC area, aged 18 to 54 years. They cannot live alone during parts of the study.

Design:

Participants will be infected with a parasite that causes malaria. The parasite will be in donated blood; it will be given through an IV.

Participants will likely develop symptoms within a week after the injection. Researchers will call daily to check on their health. After about 6 days, participants will come to the NIH clinic each day for blood tests.

Participants will check in to the NIH clinic around 10 days after the injection. They will stay in the clinic 3 to 6 days. They will have multiple blood tests every day.

Participants will be bitten by mosquitoes up to 4 times. Cups containing mosquitoes will be held against their skin for 15 minutes.

Participants will begin taking chloroquine close to the end of their clinic stay. Chloroquine is a pill taken by mouth once or twice a day for 3 days. It is FDA-approved to treat malaria.

Participants will have follow-up visits 1 and 3 weeks after discharge.

DETAILED DESCRIPTION:
Study Description: Single-center, open-label, phase 1 study to characterize the safety and infectivity of Plasmodium vivax (P. vivax) challenge agent for induced blood-stage malaria (IBSM) in malaria-naive participants at the NIH Clinical Center (NIHCC). Challenge agent derived from a cell bank of cryopreserved blood-stage P. vivax (PvHMB-CCE001) will be administered intravenously. A minimum of 2 participants will undergo IBSM to establish initial safety and infectivity of the challenge agent (pilot group). Additional participants, totaling 10 to 50 (main group), will be enrolled to further develop the model including to evaluate growth kinetics, transmission to mosquitoes using feeding assays and assess the host response to P. vivax infection. All participants who receive challenge agent will undergo antimalarial treatment. Qualification and characterization of the IBSM model, including transmission assays in malaria na(SqrRoot) ve,

unvaccinated participants, is a requisite goal in supporting future studies to evaluate stage-specific vaccines (transmission blocking

vaccines (TBVs) and blood stage vaccines (BSVs)) using the model.

Challenge agent derived from bank PvHMB-CCE001 will be assessed first in a pilot group of at least 2 participants, then subsequently in a main group with participants receiving inoculations in cohorts of up to 10 individuals based on logistical considerations including the capacity of clinic resources. The dose of the challenge agent may be adjusted if needed to generate reliable IBSM.

Objectives:

* Primary Objective

  --To assess the safety of the P. vivax IBSM model following inoculation of healthy participants.
* Secondary Objectives

  * To establish an appropriate challenge agent dose for use in P. vivax IBSM studies.
  * To evaluate transmission of P. vivax to vector mosquitoes in the IBSM model by mosquito feeding assays.
  * To establish a dataset that may be used as a historical control in future interventional IBSM transmission studies.
* Exploratory Objectives

  * To further characterize blood and sexual stage parasite growth profiles following blood-stage P. vivax challenge and treatment.
  * To assess host responses to P. vivax IBSM.
  * To optimize mosquito infectivity in feeding assays, and study human to mosquito transmission and generate mosquito stages of the parasite.
  * To establish a supply of P. vivax infected blood.

Endpoints:

* Primary Endpoint

  --Incidence and severity of local and systemic adverse events (AEs) or serious adverse events (SAEs).
* Secondary Endpoints

  * A suitable dose of challenge agent that generates parasitemia in a reliable and timely manner as determined by the investigator.
  * Transmission of P. vivax to Anopheles spp. using mosquito feeding assays including direct feeding assays and/or membrane feeding assays as determined by the detection of oocysts following midgut dissection. Additional optional measures may include salivary gland dissection or detection by molecular methods.
  * Demonstration of transmission in mosquito feeding assays among a requisite number of participants.
* Exploratory Endpoints

  * Asexual blood-stage and sexual stage parasite growth profiles by quantitative polymerase chain reaction (qPCR) and/or microscopy.
  * Antibody responses: Antibody levels elicited following IBSM as measured by enzyme-linked immunosorbent assay (ELISA) (e.g., antibodies against Pvs230, Pvs25, Pvs44/45 sexual stage antigens, or PvMSP3, MSP9, and AMA1 asexual stage antigens), cellular responses, biomarkers, and transcriptional profiling at various timepoints.
  * Collection of gametocyte-containing blood and study in mosquito transmission assays.
  * Collection of P. vivax-containing blood from participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a participant to undergo IBSM:

1. Age >=18 and <=54 years.
2. RBCs positive for Duffy antigen/chemokine receptor.
3. Malaria comprehension exam passed prior to study activities.
4. Suitable accommodation and reliable access to the NIHCC for the duration of the study in the opinion of the investigator.
5. Persons of childbearing potential must be willing to use reliable contraception from 28 days prior to challenge agent administration to the end of study.
6. Signing of the informed consent form.
7. Agreement to not live alone from challenge agent administration until the completion of antimalarial treatment.
8. Agreement to long-term storage of study samples for future research.

EXCLUSION CRITERIA:

A participant will be excluded from participating in this trial if any 1 of the following criteria is fulfilled:

1. Planned travel to a P. vivax-endemic area during the study period (see https://www.cdc.gov/malaria/travelers/country_table/a.html).
2. History of travel to or residence in a P. vivax malaria-endemic region for more than 2 weeks during the past 2 years.
3. Prior confirmed P. vivax malaria diagnosis or clinical history consistent with likely P. vivax infection. At the investigator's discretion, participants may be enrolled if the exposure was remote, e.g., > 5 years ago.
4. Poor peripheral venous access, at the discretion of the investigator.
5. For persons of childbearing potential:

   1. Currently pregnant or breastfeeding, or planning on becoming pregnant or breastfeeding until the end of study.
   2. Rh blood group negative.
6. Being a current or former study team member or clinical trial staff with direct involvement of the trial, or being an employee supervised by a study team member.
7. Unwillingness to defer blood donations for at least 3 years.
8. Use of any of the following within the specified periods:

   1. Investigational P. vivax vaccine within the last 2 years.
   2. Malaria chemoprophylaxis within 3 months of Day 0.
   3. Chronic systemic immunosuppressive medications (>14 days) within 6 months (e.g., cytotoxic medications, adrenocorticotrophic hormone, or oral/parental corticosteroids equivalent to >0.5 mg/kg/day of prednisone). Corticosteroid nasal spray for allergic rhinitis and topical corticosteroids for mild, uncomplicated dermatitis are allowed.
   4. Prior receipt of packed red cells or other blood products or immunoglobulins within the previous 6 months.
   5. Systemic antibiotics or medications with potential antimalarial effects less than 28 days before Day 0 (e.g., clindamycin, chloroquine, benzodiazepines, tetracycline, azithromycin, or doxycycline).
   6. Investigational product or vaccine less than 28 days before Day 0.
   7. Receipt of any vaccination less than 28 days before Day 0.
   8. Current or planned use of medications known to significantly prolong the QT interval or otherwise interfere with study agents.
   9. Smoking more than 5 cigarettes or equivalent per day and unable to stop smoking for the duration of admission. Participants may smoke up to 5 cigarettes or equivalent per day for the rest of the study (by attestation).
   10. History of alcohol use disorder (exceptions may be made at the investigator's discretion if they have completed treatment or are otherwise currently abstinent) or refusal to agree to refrain from drinking from the day of the challenge agent inoculation until completion of their antimalarial course.
9. Clinically significant medical condition, physical examination findings, other clinically significant abnormal laboratory results, or past medical history including:

   1. Immunodeficiency including asplenia or functional asplenia or significant autoimmune disease.
   2. Retinal disease, visual field changes, psoriasis, porphyria, or known allergy to chloroquine or artemether/lumefantrine.
   3. Cardiac disease including >10 percent cardiovascular risk as determined by the non-laboratory method or an abnormal EKG demonstrating a corrected QT interval by Fridericia's formula of >450 msec or other concerning arrhythmia.
   4. Any other medical condition that may have significant implications for current health status and participation in the study, in the opinion of the investigator.
10. History of a severe reaction to arthropod bites, or history of anaphylaxis or severe unexpected allergy to any substance.
11. Screening blood test or urinalysis laboratory parameters outside of local lab normal range (including infectious serologies). Participants may be included at the investigator's discretion for "not clinically significant" values outside of normal range.
12. Any other finding that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent, or increase the risk of having an adverse outcome from participating in the study.

Participants who are determined ineligible to participate for any of the reasons above may be rescreened for eligibility at a later time when the disqualifying condition may be resolved.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-11-26 (Estimated); Study Completion 2027-11-26 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of the P. vivax IBSM model following inoculation of healthy participants. | Time of inoculation with the challenge agent until at least 21 days after inpatient discharge
  Incidence and severity of local and systemic AEs or SAEs.

SECONDARY OUTCOMES:
To establish a dataset that may be used as a historical control in future interventional IBSM studies. | From the time of inpatient admission to the time of discharge.
  Demonstration of transmission in mosquito feeding assays among a requisite number of participants.
To evaluate transmission of P. vivax to vector mosquitoes in the IBSM model by mosquito feeding assays. | From the time of inpatient admission to the time of discharge.
  Transmission of P. vivax to Anopheles spp. using mosquito feeding assays including direct feeding assays and/or membrane feeding assays as determined by the detection of oocysts following midgut dissection. Additional optional measures may include salivary gland dissection or detection by molecular methods.
To establish an appropriate challenge agent dose for use in P. vivax IBSM studies. | From the time of inoculation until the time of inpatient admission. Expected to be approximately day 9.
  A suitable dose of challenge agent which generates parasitemia in a reliable and timely manner as determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Joel A Goldberg, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data in an NIH-funded or approved public repository.@@@- De-identified data in another public repository.@@@- Identified data in the Biomedical Translational Research Information System (automatic for activities in the CC).@@@- De-identified or identified data with approved outside collaborators under appropriate agreements.@@@- De-identified data in publications and/or public presentations.@@@Data will be shared at the time of or shortly after publication.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001970-I.html